CLINICAL TRIAL: NCT02705573
Title: Effects of Mannitol on Delayed Graft Function After Cadaveric Renal Transplantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Samir Sljivic, Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021/2014
Record Dates: First submitted 2016-03-07; First posted 2016-03-10 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Kidney Transplantation, Mannitol
MeSH Terms: interventions — Mannitol

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mannitol 20% (Experimental): Mannitol 1g/ kg BW
  Interventions: Drug: Mannitol
- Nacl 0.9% (Placebo Comparator): NaCl 0.9% 5ml/ kg BW
  Interventions: Drug: Mannitol

INTERVENTIONS:
Drug: Mannitol — In the study, mannitol 20% with a dose of 1g / kg / BW (5 ml / kg / BW) will be compared to placebo with NaCl 0.9% in the dose of 5 ml / kg / BW. The study medication will be administered immediately before organ reperfusion. The follow-up of the study is 24 hours.

SUMMARY:
In this study we want to evaluate the effect of mannitol on postoperative renal biomarkers in patient receiving cadaveric renal transplantation. Furthermore we want to evaluate the effect of mannitol on perioperative redox status in patients receiving renal transplantation using the oxidation-reduction potentials assessed with the RedoxSYS®system.

We are planning to perform a double-blind randomized controlled trial. In the study, mannitol 20% with a dose of 1g / kg / BW (5 ml / kg / BW) will be compared to placebo with NaCl 0.9% in the dose of 5 ml / kg / BW. Patients will be randomized to receive either the mannitol or NaCl. The follow-up of the study is 24 hours. The following biomarkers will be determined befor induction of anesthesia and 24 hours after administration of study medication: CCL2, CHI3LI, GH, HGF, MMP1, MMP8, Tie2, TNF-R1, VCAM-1, KIM-1, Cystatin C, FGF23, IGFB7, NGAL and IL 18.

Furthermore we want to perform sORP and cORP before induction of anesthesia, just before bolus of mannitol, 5 min after bolus of mannitol and after operation in anesthetic recovery room.

Data will be collected, compared and published at the end of the study. It is planned to include a total of 34 patients in the study.

ELIGIBILITY:
Inclusion Criteria: all patients with end stage renal diseases -

Exclusion Criteria: Patients younger than 18 years of age or older than 80, alergy to mannitol, Pregnancy, Breast-feed

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
renal biomark | 24 hours
  The BM-panel includes the following analytes: CCL2, CHI3LI, GH, HGF, MMP1, MMP8, Tie2, TNF-R1, VCAM-1, KIM-1, Cystatin C and Endostatin. Additionally, the BM-panel can be extended for measurement of FGF23, IGFB7, NGAL and IL 18.

SECONDARY OUTCOMES:
renal function parameter | 24 hours
  creatinine, blood urea, nitrogen, urinary output, potassium
oxidation-reduction potential (ORP) of mannitol | 24 hours
  static ORP (sORP), capacity ORP (cORP)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Vienna, Vienna, Austria

REFERENCES:
- [Derived] Reiterer C, Hu K, Sljivic S, Falkner von Sonnenburg M, Fleischmann E, Kabon B. The effect of mannitol on oxidation-reduction potential in patients undergoing deceased donor renal transplantation-A randomized controlled trial. Acta Anaesthesiol Scand. 2021 Feb;65(2):162-168. doi: 10.1111/aas.13713. Epub 2020 Oct 15. PMID 32966587
- [Derived] Reiterer C, Hu K, Sljivic S, Falkner von Sonnenburg M, Fleischmann E, Kainz A, Kabon B. Mannitol and renal graft injury in patients undergoing deceased donor renal transplantation - a randomized controlled clinical trial. BMC Nephrol. 2020 Jul 28;21(1):307. doi: 10.1186/s12882-020-01961-z. PMID 32723374